CLINICAL TRIAL: NCT06960590
Title: Determining the Minimal Effective Dose of Static Stretching for Increasing Range of Motion in Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Józef Piłsudski University of Physical Education (Other)
Responsible Party: Principal Investigator, Michał Kaczorowski, Principal Investigator, Józef Piłsudski University of Physical Education
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: SKE.0030.3.2025
Record Dates: First submitted 2025-04-14; First posted 2025-05-07 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-04

CONDITIONS: Static Stretching

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Streching group (Experimental): The group performed one training session per week consisting of 2 sets of static stretching
  Interventions: Other: Training - static streching
- Control group (No Intervention): Only tests were performed in the group, no intervention was introduced

INTERVENTIONS:
Other: Training - static streching — The intervention group performed one training session per week. Each training session consisted of 2 series of static stretching of the back band. The rest time between series was 45 s. The intervention lasted 6 weeks.
  Arms: Streching group

SUMMARY:
The study is planned to be conducted in 2025. The methods used in the study are non-invasive methods. The study groups will perform 1 to 3 static stretching sessions per week. The number of series per session will be from 1 to 3. The static stretching time of the back band in the series will be from 20 s to 60 s. The total stretching time per week will be from 45 s to 135 s. The break between series will be 45 s, and the duration of the intervention will be from 6 to 8 weeks. During stretching, the subject maintains a maximum bend with straight knee joints for a specified time. Before starting the study, participants will undergo a toe-to-floor test to assess the flexibility of the back band. The test will be repeated after the intervention. The aim of the study is to determine the minimum effective dose of static stretching. Currently, anecdotal evidence suggests that this dose is 90 seconds of static stretching per week.

The study does not involve any likelihood of harm to study participants as a result of participating in the study.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years,
* No lower limb injuries, no spinal injuries and no craniocerebral injuries in the last 6 months,
* No lower limb surgeries, no spinal surgeries and no central nervous system surgeries in the last 6 months,

Exclusion Criteria:

* Age under 18 years
* Injuries to the lower limbs, spine or craniocerebral injuries within the last 6 months,
* Surgical procedures to the lower limbs, spine or surgical procedures to the central nervous system within the last 6 months,

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2025-03-25 (Actual); Primary Completion 2025-08-05 (Estimated); Study Completion 2025-08-06 (Estimated)

PRIMARY OUTCOMES:
Flexibility | From registration to completion of the study, the duration is up to 8 weeks
  Flexibility was assessed using a modified stand-and-reach test. The participants stood with their feet shoulder-width apart and knees fully extended, then performed a forward bend, reaching as far as possible while maintaining straight legs. To measure the extent of their reach, a custom-built box was used. The box had the following dimensions: a length of 40 cm, a width of 45 cm, and a height of 35 cm. Each participant performed the test once. The same test was repeated after the 6-week intervention period to determine any improvements in flexibility.

CONTACTS AND LOCATIONS:
Locations (1):
- Józef Piłsudski Academy of Physical Education in Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shadmehr A, Hadian MR, Naiemi SS, Jalaie S. Hamstring flexibility in young women following passive stretch and muscle energy technique. J Back Musculoskelet Rehabil. 2009;22(3):143-8. doi: 10.3233/BMR-2009-0227. PMID 20023343
- [Background] Thomas E, Bianco A, Paoli A, Palma A. The Relation Between Stretching Typology and Stretching Duration: The Effects on Range of Motion. Int J Sports Med. 2018 Apr;39(4):243-254. doi: 10.1055/s-0044-101146. Epub 2018 Mar 5. PMID 29506306
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/29506306/